CLINICAL TRIAL: NCT02214134
Title: SPECTAlung: Screening Patients With Thoracic Tumors for Efficient Clinical Trial Access
Acronym: SPECTAlung
Status: Completed | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1335-LCG-PBG
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Any Stage of Lung Cancer (Any Histotype); Any Stage of Malignant Pleural Mesothelioma; Any Stage of Any Thymic Malignancy
Keywords: Lung cancer; Malignant pleural mesothelioma; Thymic malignancy; Biomarkers; Screening
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — FFPE blocks of tumour tissue Blood samples Pleural effusion samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Lung cancer: Patients with diagnosis of lung cancer at any stage
  Interventions: Genetic: Tumour markers testing
- Malignant pleural mesothelioma: Patients with diagnosis of malignant pleural mesothelioma at any stage
  Interventions: Genetic: Tumour markers testing
- Thymic malignancy: Patients with diagnosis of thymic malignancy at any stage
  Interventions: Genetic: Tumour markers testing

INTERVENTIONS:
Genetic: Tumour markers testing

SUMMARY:
SPECTAlung is a program aiming at screening patients with thoracic tumors to identify the molecular characteristics of their disease. The thoracic tumors include lung cancer, malignant pleural mesothelioma, thymoma or thymic carcinoma at any stage. Once the molecular characteristics are identified, there might be the possibility to offer these patients access to targeted clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed lung cancer, MPM, thymoma or thymic carcinoma at any stage;
* Mandatory availability of adequate Human Biological Material (HBM): FFPE tissue sample from the primary tumor, recurrent tumor, metastasis, obtained at the time of primary surgery or biopsy; minimal amount requested is detailed in the HBM guidelines; inclusion of samples taken at any recurrence diagnosed during follow-up is strongly encouraged but optional;
* Centrally performed confirmation of tumor tissue adequacy in terms of quality/ quantity for central screening;
* Age ≥ 18 years;
* At least three months life-expectancy;
* Written informed consent according to ICH/GCP and national/local regulations.

Exclusion Criteria:

* Any active malignancy, except pT1-2 prostatic cancer Gleason score < 6, non melanomatous skin cancer or carcinoma in situ of the cervix, in the 5 years before study entry;
* Active hepatitis B/C or HIV;
* Any secondary malignancy;
* Any severe organ dysfunction or other comorbidities that may prevent the inclusion into clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically confirmed lung cancer, MPM, thymoma or thymic carcinoma at any stage.
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with thoracic malignancy (lung cancer, MPM and thymic malignancies) screened and efficiently allocated to biomarker-driven clinical trials. | 5 years

SECONDARY OUTCOMES:
Number of patients for whom the description of the biomarkers and correlation to clinical/pathological characteristics can be performed. | 5 years
Number of exploratory/future research projects developped | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Besse, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (17):
- Belgium (3):
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- France (4):
  - CHU de Lyon - Hopital Louis Pradel, Lyon
  - Assistance Publique - Hopitaux de Marseille - Hopital Nord, Marseille
  - CHU Toulouse - Hopital Larrey, Toulouse
  - Gustave Roussy Cancer Campus, Villejuif
- St. James's Hospital, Dublin, Ireland
- Ospedale S. Luigi Gonzaga - Universita Di Torino, Torino, Italy
- Medical University Of Gdansk, Gdansk, Poland
- University Clinic Golnik, Golnik, Slovenia
- Spain (2):
  - Hospital General Vall D'Hebron, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
- Centre Hospitalier Universitaire Vaudois - Lausanne, Lausanne, Switzerland
- United Kingdom (3):
  - Royal Marsden Hospital - Kingston Hospital, Kingston upon Thames
  - Royal Marsden Hospital - Chelsea, London, London
  - Royal Marsden Hospital - Sutton, Surrey, Sutton